CLINICAL TRIAL: NCT03098043
Title: Post-Static Cold Storage Hypothermic Oxygenated Perfusion in Bergamo Liver Transplant Program: a Prospective Observational Study
Brief Title: Post-Static Cold Storage Hypothermic Oxygenated Perfusion in Bergamo Liver Transplant Program
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Papa Giovanni XXIII Hospital (Other)
Responsible Party: Principal Investigator, Stefania Camagni, MD, Papa Giovanni XXIII Hospital
Other Study IDs: Post-SCS Liver HOPE Bg
Record Dates: First submitted 2017-03-26; First posted 2017-03-31 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Liver Transplantation
Keywords: Hypothermic machine perfusion; Donation after circulatory death; Extended criteria liver grafts

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In light of the widespread organ shortage, dynamic preservation by means of Machine Perfusion (MP) has been proposed as a strategy to increase the pool of suitable grafts for liver transplantation. Reproducing more physiological conditions than traditional Static Cold Storage (SCS), MP may allow a better preservation and evaluation and perhaps even the resuscitation of high risk grafts. As a consequence, unnecessary discard of organs could be avoided and quality and safety of transplantation could be improved as well.

Hypothermic MP (HMP) seems to reduce ischemia-reperfusion injury. In fact, hypothermia slows down the metabolic rate and the oxygenation of the perfusate leads to re-synthesis of Adenosine TriPhosphate (ATP), which results in the restoration of cellular energy.

Four series about the use of HMP in the clinical setting has been published so far. They all report acceptable outcomes after transplantation of human liver grafts from extended criteria Brain Dead Donors (BDD) and from Donation after Circulatory Death (DCD) donors preserved by HMP, thus proving its feasibility and safety. The efficacy of HMP, instead, is still under investigation in a phase II randomized trial.

This is an observational, prospective, monocentric study aiming at verifying the feasibility and safety of post-SCS Hypothermic Oxygenated PErfusion (HOPE) in the setting of our liver transplant program. Extended criteria grafts from BDD and grafts from DCD donors will be preserved by post-SCS HOPE prior to transplantation. The recipients of these grafts will be followed-up for at least 1 year.

DETAILED DESCRIPTION:
This is an observational, prospective, monocentric study aiming at verifying the feasibility and safety of post-SCS HOPE in the setting of our liver transplant program.

20 consecutive patients with written informed consent will be enrolled. They will be transplanted with grafts from extended criteria BDD or from DCD donors preserved by post-SCS HOPE.

The HOPE procedure will be performed in our operating room after regular procurement, transport and back-table preparation. University of Wisconsin Machine Perfusion Solution (UW-MPS) will be used. Two pumps will provide dual pressure-controlled perfusion through the portal vein and the hepatic artery. Portal flow will be continuous and will be adjusted to keep portal pressure below 5 mmHg. Instead, arterial flow will be pulsatile and will be regulated to maintain arterial pressure between 25 mmHg and 30 mmHg. The perfusate will be oxygenated with the goal of a partial Pressure of Oxygen (PO2) of 50-70 kilopascal. The perfusate temperature will be kept between 4°C and 12°C by a heat exchanger. pH, PO2 and partial Pressure of Carbon Dioxide (PCO2) of the perfusate pumped to the graft and drained from the vena cava will be monitored. HOPE will be maintained for 3 to 4 hours.

Patients will be followed-up for at least 1 year according to a scheduled timetable.

Data about HOPE and transplant procedure, about donors and recipients' characteristics and about patients' follow-up will be collected in a dedicated electronic Case Report Form (eCRF) according to Good Clinical Practice.

ELIGIBILITY:
Grafts inclusion criteria:

* extended criteria BDD with a mix of the following: age ≥70 years, liver macrosteatosis ≥35%, anti-Hepatitis C Virus (HCV) positivity, Hepatitis B surface Antigen (HBsAg) positivity, hemodynamic instability
* DCD donors category IVB (on ExtraCorporeal Membrane Oxygenation (ECMO) support) with a mix of the above-mentioned characteristics and/or with undetermined hepatocellular necrosis
* DCD donors category I-IVA on normothermic regional ECMO support
* different donors characteristics from the above-mentioned ones but organisational set-up including prolonged total ischemic time.

Grafts exclusion criteria: living donors.

Recipients' inclusion criteria:

* liver transplant candidates who are going to be transplanted with a graft preserved by post-SCS HOPE
* liver transplant candidates who consent to participate in the study by signing the informed consent form.

Recipients' exclusion criteria:

* liver transplant candidates who are going to be transplanted with a graft preserved by SCS
* liver transplant candidates who are going to be transplanted with a graft preserved by post-SCS HOPE but refuse consent for their participation in the study.

Ages: 30 Days to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the patients on the waiting list for liver transplantation at Bergamo transplant centre, except for those who are candidates to combined en bloc liver and pancreas transplantation
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2017-11-05 (Actual); Primary Completion 2021-12-03 (Estimated); Study Completion 2021-12-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of early allograft dysfunction (safety endpoint) | Post-operative day 7
  Occurrence of one or more of the following: bilirubin >170 µmol/L on Post-Operative Day (POD) 7, International Normalized Ratio (INR) >1,6 on POD 7, Alanine AminoTransferase (ALT) peak >2000 U/L within the first post-operative week

SECONDARY OUTCOMES:
Rate of complications grade ≥IIIa | 1 year after transplantation
  Dindo-Clavien classification of surgical complications
Incidence of ischemic cholangiopathy | 6 months after transplantation
  Radiological or endoscopic diagnosis of unifocal or multifocal intrahepatic strictures in the absence of any arterial complication
Length of intensive care unit and hospital stay | 1 year after transplantation
  Length of intensive care unit and hospital stay after transplantation (days)
30-day patient survival | Post-operative day 30
  Patient survival rate 30 days after transplantation
30-day graft survival | Post-operative day 30
  Graft survival rate 30 days after transplantation
1-year patient survival | 1 year after transplantation
  Patient survival rate 1 year after transplantation
1-year graft survival | 1 year after transplantation
  Graft survival rate 1 year after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Stefania Camagni, MD, Principal Investigator — Papa Giovanni XXIII Hospital; Michele Colledan, MD, Study Director — Papa Giovanni XXIII Hospital
Locations (1):
- Papa Giovanni XXIII Hospital, Bergamo, Italy

IPD SHARING:
Plan to Share IPD: No